CLINICAL TRIAL: NCT04134143
Title: An Open-Label, Prospective, Safety, and Tolerability Study of ExpressGraft- C9T1 Skin Tissue in the Treatment of Diabetic Foot Ulcers
Brief Title: Multiple Applications of ExpressGraft-C9T1 Skin Tissue as a Treatment for Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision - not related to product quality or safety concerns
Sponsor: Stratatech, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C9T12015 (Extended)
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Diabetes; Diabetic Foot Ulcer; Non-healing Wound
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Cohort 2 will begin when the study starts, and after the safety monitoring board approves progression to the next cohort, Cohort 3 will begin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: One Application (Experimental): Participants enrolled in Cohort 1 received one application of experimental skin tissue during the first part of this trial (NCT02657876)
  Interventions: Biological: ExpressGraft-C9T1 Skin Tissue
- Cohort 2: Up to Five Applications (Experimental): Participants enrolled in Cohort 2 may receive up to 5 applications of experimental skin tissue as required for wound healing
  Interventions: Biological: ExpressGraft-C9T1 Skin Tissue
- Cohort 3: Up to Ten Applications (Experimental): Participants enrolled in Cohort 3 may receive up to 10 applications of experimental skin tissue as required for wound healing
  Interventions: Biological: ExpressGraft-C9T1 Skin Tissue

INTERVENTIONS:
Biological: ExpressGraft-C9T1 Skin Tissue — A round patch of experimental skin tissue that the doctor applies over the ulcer
  Other Names: Experimental skin tissue

SUMMARY:
Some people with diabetes get foot ulcers that do not heal. These ulcers can get infected and cause other medical problems.

Five patients with these foot ulcers volunteered to participate in the first part of this study (C9T12015, NCT02657876). They are called Cohort 1 in this registration. Cohort 1 received one application (piece) of an experimental skin tissue to make sure it was safe.

This study will extend the safety test of the experimental skin tissue. It will find out if it is safe to use more than once to cover non-healing ulcers.

This extension will include two more groups, Cohort 2 and Cohort 3. Cohort 2 may get up to 5 applications. Cohort 3 may get up to 10 applications. The number of applications will depend on how well the wound is healing.

Participants will be in the study up to one year.

ELIGIBILITY:
Volunteers will be consented. Then there will be a run-in period for the doctor to run some tests. If the tests show the study would be good for the patient, the doctor will enroll them as participants in the trial.

Inclusion Criteria:

To be considered for inclusion, a participant:

* Agrees to practice birth control for the duration of the study
* Has documented Type 1 or Type 2 diabetes and an HbA1C score of 10 or below
* Has protocol-defined sufficient blood pressure and flow to the foot
* Has stable medications for 2 weeks before treatment (other than diabetes medications or antibiotics)
* Is able and willing to attend scheduled visits and comply with study procedures
* If a smoker, agrees to try quitting and will accept counseling for it (Cohorts 2 and 3 only)
* Has documented informed consent for study enrollment
* Has had an uninfected, appropriately-sized diabetic ulcer on the foot for at least 4 weeks but not more than 1 year

Exclusion Criteria:

The doctor may not consider for inclusion a participant who:

* Is pregnant, nursing, or a prisoner
* Has had osteomyelitis in the foot with the ulcer in the last 30 days
* Has a history of poor compliance
* Has received drugs or therapies not allowed per protocol
* Has used an investigational product within the last 60 days
* Has ever received therapy for the study ulcer with any cell and/or tissue product (CTP)
* Has a study ulcer in a condition not appropriate for the study
* Has a medical condition or history that, per protocol or in the opinion of the study doctor, might put the safety of the participant in danger

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events at Week 12 | at Week 12
  Clinically significant vital signs, infection, blood chemistry, hematology and immunological evaluations are recorded as adverse events
Number of participants with adverse events through study completion | at approximately 12 months
  Clinically significant vital signs, infection, blood chemistry, hematology and immunological evaluations are recorded as adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Stratatech, a Mallinckrodt Company
Locations (4):
- United States (4):
  - Titan Clinical Research, Phoenix, Arizona
  - Limb Preservation Platform, Inc., Fresno, California
  - Center For Clinical Resarch, San Francisco, California
  - Center for Advanced Research & Education, Gainesville, Georgia

IPD SHARING:
Plan to Share IPD: No